CLINICAL TRIAL: NCT04464304
Title: Virtual Reality for Postoperative Pain Management After Head and Neck Surgery: A Randomized Controlled Trial
Brief Title: Virtual Reality for Postoperative Pain Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Ryan Li, MD, Assistant Professor of Otolaryngology - Head and Neck Surgery, Division of Head and Neck Surgery, School of Medicine, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 00020777
Record Dates: First submitted 2020-07-06; First posted 2020-07-09 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Surgery; Pain, Postoperative; Incision; Otolaryngological Disease
Keywords: Virtual Reality
MeSH Terms: conditions — Pain, Postoperative; Surgical Wound; Otorhinolaryngologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (Active Comparator): Patients will be provided with a commercially-available VR device for use up to 15 minutes at bedside.
  Interventions: Device: Virtual Reality (Oculus Quest)
- Smartphone (Sham Comparator): Patients will be provided with a commercially-available smartphone device for use up to 15 minutes at bedside.
  Interventions: Device: Smartphone

INTERVENTIONS:
Device: Smartphone — Patients will participate in a similar game to the VR cohort, but will use a smartphone device.
  Arms: Smartphone
Device: Virtual Reality (Oculus Quest) — Patients will participate in a game using VR.
  Arms: Virtual Reality

SUMMARY:
This trial studies an active virtual reality (VR) experience as a means for non-pharmacologic postoperative pain management among patients after head and neck surgery. Investigators will assess differences in pain scores, analgesic use, and subjective patient experiences between patients participating in a VR activity and patients participating in the same activity using a smartphone.

DETAILED DESCRIPTION:
Management of postoperative pain after head and neck surgery is complex, and has received increased attention to improve patient recovery and quality of life. Narcotic analgesics are frequently utilized in postoperative pain management, but these have risks including nausea, sedation, constipation, and dependence. Multimodal analgesia can reduce narcotic use and improve recovery, but medical comorbidities may contraindicate the use of certain medications. Non-pharmacologic measures for postoperative pain control may provide novel and cost-effective strategies to confront this complex issue.

Patients undergoing head and neck surgery will be randomly allocated to participate in an immersive experience in VR, or to participate in a similar experience on a two-dimensional screen using a smartphone.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone head and neck surgery with an average pain score of 3 or greater out of 10 during the 24 hours preceding the screening
* Are able to provide informed consent
* Are not in the intensive care unit (ICU)

Exclusion Criteria:

* Symptoms concerning for an active respiratory infection including fever, cough, and shortness of breath or confirmed respiratory infection
* Active eye discharge
* Active nausea or vomiting
* History of seizure, epilepsy, or hypersensitivity to flashing light
* History of motion sickness or vertigo
* Have wound dressings on the head or neck that prevent comfortable and safe use of the virtual reality headset

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-07-11 (Actual); Primary Completion 2021-10-20 (Actual); Study Completion 2021-10-20 (Actual)

PRIMARY OUTCOMES:
Change in patient-reported pain scores | Up to 4 hours after intervention use
  Pain scores will be obtained using an 11-point Numeric Rating Scale (NRS) prior to each intervention, immediately after the intervention, and then hourly up to 4 hours after the intervention to assess changes in pain scores after each intervention. A score of 0 signifies no pain, and a score of 10 signifies the highest severity of pain.

SECONDARY OUTCOMES:
Opioid usage | Average 24 hours after intervention use
  Opioid use after intervention will be documented, measured in average morphine milligram equivalents (MME).
Patient experience | Up to 4 hours after intervention use
  Patients will complete a short survey at the completion of their participation in the study evaluating their audiovisual experience using a 5-point Likert scale, with responses ranging from "1 = Strongly Disagree" to "5 = Strongly Agree."

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Li, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pandrangi VC, Shah SN, Bruening JD, Wax MK, Clayburgh D, Andersen PE, Li RJ. Effect of Virtual Reality on Pain Management and Opioid Use Among Hospitalized Patients After Head and Neck Surgery: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2022 Aug 1;148(8):724-730. doi: 10.1001/jamaoto.2022.1121. PMID 35679057